CLINICAL TRIAL: NCT04758689
Title: Laser Acupuncture in Rheumatoid Arthritis Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, A. Sedky, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/002-2021
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Lasers; Exercise; Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser acupuncture and aerobic exercise (Experimental)
  Interventions: Combination Product: Laser, exercise, and methotrexate
- Aerobic exercise (Experimental)
  Interventions: Combination Product: Exercise, and methotrexate

INTERVENTIONS:
Combination Product: Laser, exercise, and methotrexate — Laser therapy at acupuncture points, aerobic exercise, and methotrexate
  Arms: Laser acupuncture and aerobic exercise
Combination Product: Exercise, and methotrexate — Aerobic exercise, and methotrexate
  Arms: Aerobic exercise

SUMMARY:
Studying the effect of laser acupuncture on geriatric patients with rheumatoid arthritis

ELIGIBILITY:
Inclusion Criteria:

* Patients referred from physician (immunologist) diagnosed with rheumatoid arthritis.

Exclusion Criteria:

* Patients having the disease overlapping with other connective tissue diseases, such as systematic lupus erythromatosus and systematic sclerosis.
* History of malignancies.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Interleukin 6 (IL-6) | Baseline
  interleukin 6
Interleukin 6 (IL-6) | 4 weeks
  interleukin 6
Malondialdehyde (MDA) | Baseline
  malondialdehyde
Malondialdehyde (MDA) | 4 weeks
  malondialdehyde
Adenosine Triphosphate (ATP) | Baseline
  adenosine triphosphate
Adenosine Triphosphate (ATP) | 4 weeks
  adenosine triphosphate
C-Reactive Protein (CRP) | Baseline
  C-reactive protein
C-Reactive Protein (CRP) | 4 weeks
  C-reactive protein

SECONDARY OUTCOMES:
Rheumatoid Arthritis Quality of Life (RAQoL) | Baseline
  rheumatoid arthritis quality of life
Rheumatoid Arthritis Quality of Life (RAQoL) | 4 weeks
  rheumatoid arthritis quality of life
Health Assessment Questionnaire (HAQ) | Baseline
  health assessment questionnaire
Health Assessment Questionnaire (HAQ) | 4 weeks
  health assessment questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- A. Sedky, Cairo, Egypt

REFERENCES:
- [Derived] Adly AS, Adly AS, Adly MS. Effects of laser acupuncture tele-therapy for rheumatoid arthritis elderly patients. Lasers Med Sci. 2022 Feb;37(1):499-504. doi: 10.1007/s10103-021-03287-0. Epub 2021 Mar 19. PMID 33738615